CLINICAL TRIAL: NCT01648699
Title: Study on the Effectiveness and Safety of OROS Hydromorphone in Pain Management Among Patients With Cancer Pain
Brief Title: Safety and Efficacy Study of Osmotic Release Oral System (OROS) Hydromorphone in Participants With Cancer Pain
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: the study was stopped due to non-availability of 4mg
Sponsor: Janssen Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR016351; 42801PAI4008
Record Dates: First submitted 2012-07-20; First posted 2012-07-24 (Estimated); Results first posted 2013-10-11 (Estimated); Last update posted 2013-10-11 (Estimated); Status verified 2013-10

CONDITIONS: Pain
Keywords: Pain; Cancer; Osmotic Release Oral System; OROS Hydromorphone; Jurnista
MeSH Terms: conditions — Pain; Neoplasms | interventions — Hydromorphone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Osmotic Release Oral System (OROS) Hydromorphone (Experimental): OROS Hydromorphone will be administered as either 8, 12, 16, 20, 24, 32, 36 or 40 mg oral tablet once daily in the morning. For all participants, 24-hour stable opioid dose (of either morphine or oxycodone) will be converted to a single daily dose of OROS hydromorphone using standard equi-analgesic ratios and dose will be increased if needed, but not more than 40 mg and not more frequently than every two days. The study drug will be administered up to 28 days.
  Interventions: Drug: Osmotic Release Oral System (OROS) hydromorphone

INTERVENTIONS:
Drug: Osmotic Release Oral System (OROS) hydromorphone — OROS Hydromorphone will be administered as either 8, 12, 16, 20, 24, 32, 36 or 40 mg oral tablet once daily in the morning. For all participants, 24-hour stable opioid dose (of either morphine or oxycodone) will be converted to a single daily dose of OROS hydromorphone using standard equi-analgesic ratios and dose will be increased if needed, but not more than 40 mg and not more frequently than every two days. The study drug will be administered up to 28 days.
  Other Names: Jumista

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of Osmotic Release Oral System (OROS) hydromorphone using standardized conversion from prior opioid therapy among participants with cancer pain.

DETAILED DESCRIPTION:
This is a prospective (study following participants forward in time), open-label (all people know the identity of the intervention), single-arm, multi-center (conducted in more than one center) study to evaluate the effectiveness and safety of stable dose of OROS hydromorphone among participants with cancer pain. The duration of this study will be 28 days and will include visits at: Day 0 (Baseline), Day 7, 14 and 28. The OROS hydromorphone will be administered orally for 28 days and dose titration (incremental increase in drug dosage to a level that provides the optimal therapeutic effect) will be done every two days upon administration of dose. Rescue medication (a medication intended to relieve symptoms immediately) of morphine will be permitted throughout the study duration. Efficacy of the participants will primarily be evaluated by Brief Pain Inventory score. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant with histological confirmed malignancy
* Participant on stable morphine or 25 milligram oxycodone dose equivalent per day. Stable dose is defined as no dose change for 3 consecutive days and does not require more than 3 doses of rescue medication per day
* Life expectancy of at least 3 months
* Negative urine pregnancy test
* Participants with signed informed consent

Exclusion Criteria:

* Participant intolerant or hypersensitive to hydromorphone or other opioid agonist
* Participant with unstable medical condition
* Participant with renal dysfunction and liver dysfunction
* Participant dependence to opiates
* Inability to take oral medication

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica Clinical Trial, Study Director — Janssen Pharmaceutica

RESULTS

PARTICIPANT FLOW:
Groups:
- Osmotic Release Oral System (OROS) Hydromorphone: Osmotic Release Oral System (OROS) Hydromorphone was administered as either 8, 12, 16, 20, 24, 32, 36 or 40 milligram (mg) oral tablet once daily in the morning. For all participants, 24-hour stable opioid dose (of either morphine or oxycodone) was converted to a single daily dose of OROS hydromorphone using standard equi-analgesic ratios and was increased if needed, but not more frequently than every two days and not more than 40 mg. The study drug was administered up to 28 days.
Period: Overall Study
Arm/Group | Osmotic Release Oral System (OROS) Hydromorphone
Started | 20
Completed | 15
Not Completed | 5
Not completed — Death | 1
Not completed — Lost to Follow-up | 2
Not completed — Unspecified/unable to complete 4 visits | 2

BASELINE CHARACTERISTICS:
Arm/Group | Osmotic Release Oral System (OROS) Hydromorphone
Number analyzed (Participants) | 20
Age Continuous [Mean (Standard Deviation); unit: Years] | 50.35 (11.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Brief Pain Inventory (BPI) Average Score at Baseline
Description: The Brief Pain Inventory (BPI) assesses the severity of pain and the impact of pain on daily functions (interference items). The severity items are scored from 0=no pain and 10=pain as bad as you can imagine. The interference items are scored from 0=no interference and 10=interferes completely.
Time Frame: Baseline
Population: Intent-to-treat (ITT) population included all participants who received at least one dose of study medication at Baseline.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- OROS Hydromorphone 8 Milligram (mg): OROS Hydromorphone was administered as 8 mg oral tablet once daily in the morning. For all participants, 24-hour stable opioid dose (of either morphine or oxycodone) was converted to a single daily dose of OROS hydromorphone using standard equi-analgesic ratios and was increased if needed, but not more frequently than every two days. The study drug was administered up to 28 days.
- OROS Hydromorphone 12 mg: OROS Hydromorphone was administered as 12 mg oral tablet once daily in the morning. For all participants, 24-hour stable opioid dose (of either morphine or oxycodone) was converted to a single daily dose of OROS hydromorphone using standard equi-analgesic ratios and was increased if needed, but not more frequently than every two days. The study drug was administered up to 28 days.
- OROS Hydromorphone 16 mg: OROS Hydromorphone was administered as 16 mg oral tablet once daily in the morning. For all participants, 24-hour stable opioid dose (of either morphine or oxycodone) was converted to a single daily dose of OROS hydromorphone using standard equi-analgesic ratios and was increased if needed, but not more frequently than every two days. The study drug was administered up to 28 days.
- OROS Hydromorphone 20 mg: OROS Hydromorphone was administered as 20 mg oral tablet once daily in the morning. For all participants, 24-hour stable opioid dose (of either morphine or oxycodone) was converted to a single daily dose of OROS hydromorphone using standard equi-analgesic ratios and was increased if needed, but not more frequently than every two days. The study drug was administered up to 28 days.
- OROS Hydromorphone 24 mg: OROS Hydromorphone was administered as 24 mg oral tablet once daily in the morning. For all participants, 24-hour stable opioid dose (of either morphine or oxycodone) was converted to a single daily dose of OROS hydromorphone using standard equi-analgesic ratios and was increased if needed, but not more frequently than every two days. The study drug was administered up to 28 days.
- OROS Hydromorphone 32 mg: OROS Hydromorphone was administered as 32 mg oral tablet once daily in the morning. For all participants, 24-hour stable opioid dose (of either morphine or oxycodone) was converted to a single daily dose of OROS hydromorphone using standard equi-analgesic ratios and was increased if needed, but not more frequently than every two days. The study drug was administered up to 28 days.
- OROS Hydromorphone 36 mg: OROS Hydromorphone was administered as 36 mg oral tablet once daily in the morning. For all participants, 24-hour stable opioid dose (of either morphine or oxycodone) was converted to a single daily dose of OROS hydromorphone using standard equi-analgesic ratios and was increased if needed, but not more frequently than every two days. The study drug was administered up to 28 days.
Arm/Group | OROS Hydromorphone 8 Milligram (mg) | OROS Hydromorphone 12 mg | OROS Hydromorphone 16 mg | OROS Hydromorphone 20 mg | OROS Hydromorphone 24 mg | OROS Hydromorphone 32 mg | OROS Hydromorphone 36 mg
Number analyzed (Participants) | 5 | 6 | 3 | 2 | 1 | 1 | 2
Units on a scale
  Severity item: Worst pain in last 24 hours | 7.40 (1.82) | 6.50 (3.45) | 4.00 (4.00) | 10.00 (0.00) | 2.00 (0.00) | 8.0 (0.00) | 5.0 (2.83)
  Severity item: Least pain in last 24 hours | 2.60 (2.70) | 1.00 (1.67) | 1.00 (1.73) | 3.00 (1.41) | 0.00 (0.00) | 3.0 (0.00) | 3.5 (4.95)
  Severity item: Average pain | 5.50 (2.78) | 2.50 (1.97) | 3.00 (2.65) | 5.50 (0.71) | 1.00 (0.00) | 5.0 (0.00) | 3.5 (4.95)
  Severity item: Pain right now | 4.60 (4.03) | 2.00 (2.28) | 2.67 (3.06) | 7.00 (4.24) | 4.00 (0.00) | 3.0 (0.00) | 5.0 (4.24)
  Interference item: General activity | 6.20 (4.27) | 4.50 (3.39) | 4.33 (3.79) | 6.50 (2.12) | 0.00 (0.00) | 8.0 (0.00) | 7.0 (1.41)
  Interference item: Mood | 7.00 (1.87) | 3.00 (2.37) | 5.33 (4.73) | 6.00 (1.41) | 5.00 (0.00) | 7.00 (0.00) | 6.00 (1.41)
  Interference item: Walking ability | 7.40 (1.82) | 4.17 (4.22) | 5.33 (4.62) | 8.00 (2.83) | 3.00 (0.00) | 7.00 (0.00) | 6.50 (0.71)
  Interference item: Normal work | 5.00 (3.61) | 5.83 (4.12) | 6.33 (5.51) | 9.00 (1.41) | 0.00 (0.00) | 9.00 (0.00) | 9.00 (1.41)
  Interference item: Relationships with other people | 3.00 (3.74) | 2.33 (3.88) | 3.33 (4.16) | 6.50 (4.95) | 8.00 (0.00) | 9.00 (0.00) | 4.50 (4.95)
  Interference item: Sleep | 6.80 (3.83) | 2.33 (3.20) | 2.67 (4.62) | 8.00 (0.00) | 0.00 (0.00) | 5.00 (0.00) | 4.50 (4.95)
  Interference item: Enjoyment of life | 5.40 (4.51) | 3.17 (4.02) | 5.00 (4.36) | 7.50 (0.71) | 7.00 (0.00) | 8.00 (0.00) | 4.00 (5.66)

2. Primary Outcome: Brief Pain Inventory (BPI) Average Score at Day 28
Description: The BPI assesses the severity of pain and the impact of pain on daily functions (interference items). The severity items are scored from 0=no pain and 10=pain as bad as you can imagine. The interference items are scored from 0=no interference and 10=interferes completely.
Time Frame: Day 28
Population: ITT population included all participants who received at least one dose of study medication at Baseline. 'N ' (number of participants analyzed) signifies the participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- OROS Hydromorphone 40 mg: OROS Hydromorphone was administered as 40 mg oral tablet once daily in the morning. For all participants, 24-hour stable opioid dose (of either morphine or oxycodone) was converted to a single daily dose of OROS hydromorphone using standard equi-analgesic ratios and was increased if needed, but not more frequently than every two days. The study drug was administered up to 28 days.
Arm/Group | OROS Hydromorphone 8 Milligram (mg) | OROS Hydromorphone 12 mg | OROS Hydromorphone 16 mg | OROS Hydromorphone 20 mg | OROS Hydromorphone 24 mg | OROS Hydromorphone 32 mg | OROS Hydromorphone 40 mg
Number analyzed (Participants) | 1 | 5 | 1 | 2 | 1 | 3 | 1
Units on a scale
  Severity item: Worst pain in last 24 hours | 2.00 (0.00) | 3.20 (3.35) | 0.00 (0.00) | 4.00 (5.66) | 4.00 (0.00) | 7.00 (3.61) | 7.00 (0.00)
  Severity item: Least pain in last 24 hours | 0.00 (0.00) | 2.40 (3.05) | 0.00 (0.00) | 1.50 (2.12) | 0.00 (0.00) | 3.67 (4.04) | 3.00 (0.00)
  Severity item: Average pain | 2.00 (0.00) | 2.40 (3.21) | 0.00 (0.00) | 1.50 (2.12) | 0.00 (0.00) | 5.33 (3.06) | 4.00 (0.00)
  Severity item: Pain right now | 2.00 (0.00) | 1.00 (2.24) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 6.67 (4.04) | 3.00 (0.00)
  Interference item: General activity | 2.00 (0.00) | 4.20 (4.60) | 0.00 (0.00) | 5.00 (7.07) | 0.00 (0.00) | 7.33 (4.62) | 7.00 (0.00)
  Interference item: Mood | 2.00 (0.00) | 1.80 (3.03) | 0.00 (0.00) | 5.00 (7.07) | 0.00 (0.00) | 4.67 (2.89) | 7.00 (0.00)
  Interference item: Talking ability | 0.00 (0.00) | 4.00 (4.69) | 0.00 (0.00) | 5.00 (7.07) | 0.00 (0.00) | 8.00 (3.46) | 7.00 (0.00)
  Interference item: Normal work | 2.00 (0.00) | 3.20 (4.32) | 0.00 (0.00) | 5.00 (7.07) | 0.00 (0.00) | 8.00 (3.46) | 7.00 (0.00)
  Interference item: Relationships with other people | 1.00 (0.00) | 1.80 (3.49) | 0.00 (0.00) | 5.00 (7.07) | 0.00 (0.00) | 5.00 (4.58) | 5.00 (0.00)
  Interference item: Sleep | 1.00 (0.00) | 2.60 (3.44) | 0.00 (0.00) | 2.00 (2.83) | 0.00 (0.00) | 7.33 (3.06) | 5.00 (0.00)
  Interference item: Enjoyment of life | 1.00 (0.00) | 1.20 (2.17) | 0.00 (0.00) | 4.00 (5.66) | 0.00 (0.00) | 5.33 (4.04) | 5.00 (0.00)

3. Secondary Outcome: Number of Participants Given Rescue Pain Medications
Description: Rescue medication was a medication intended to relieve symptoms immediately. Rescue medication of morphine was used during the study duration and dose was set at 10-15 percent of the total daily morphine dose which ranged from 10-60 milligram.
Time Frame: Day 28
Population: as for outcome 2
Measure: Number; unit: Participants
Groups:
- OROS Hydromorphone (No Dose Indicated): OROS Hydromorphone was administered as either 8, 12, 16, 20, 24, 32, 36 or 40 mg oral tablet once daily in the morning for 28 days, as the dose was not indicated for these participants.
Arm/Group | OROS Hydromorphone 8 Milligram (mg) | OROS Hydromorphone 12 mg | OROS Hydromorphone 16 mg | OROS Hydromorphone 20 mg | OROS Hydromorphone 24 mg | OROS Hydromorphone 32 mg | OROS Hydromorphone 40 mg | OROS Hydromorphone (No Dose Indicated)
Number analyzed (Participants) | 1 | 5 | 1 | 2 | 1 | 2 | 1 | 2
Participants | 1 | 4 | 0 | 1 | 1 | 2 | 1 | 2

4. Secondary Outcome: Number of Participants With Categorical Score on Clinical Global Impression Scale as Assessed by Clinician
Description: The Clinical Global Impression (CGI) rating scale is a 7-point global assessment that measures the clinician's impression of the severity of illness exhibited by a participant, which ranges from "very much worse" to "very much improved" (as compared to Baseline).
Time Frame: Day 28
Population: ITT population included all participants who received at least one dose of study medication at Baseline. "n" signifies those participants who were evaluated for this measure at the specified time point. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: Participants
Groups:
- OROS Hydromorphone: OROS Hydromorphone was administered as either 8, 12, 16, 20, 24, 32, 36 or 40 mg oral tablet once daily in the morning. For all participants, 24-hour stable opioid dose (of either morphine or oxycodone) was converted to a single daily dose of OROS hydromorphone using standard equi-analgesic ratios and was increased if needed, but not more frequently than every two days and not more than 40 mg. The study drug was administered up to 28 days.
Arm/Group | OROS Hydromorphone
Number analyzed (Participants) | 15
Participants
  Very much improved: Day 28 (n=15) | 7
  Much improved: Day 28 (n=15) | 3
  Minimally improved: Day 28 (n=15) | 3
  No change: Day 28 (n=15) | 1
  Minimally worse: Day 28 (n=15) | 0
  Very much worse: Day 28 (n=15) | 0
  Not evaluated: Day 28 (n=15) | 1

ADVERSE EVENTS:
Time Frame: Baseline up to Day 28
Description: An adverse event is any untoward medical occurrence in a clinical study participant administered with study treatment. It can be any unfavorable and unintended sign/abnormal finding, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Arm/Group | OROS Hydromorphone
Serious Adverse Events (participants affected / at risk) | 2/20
Other Adverse Events (participants affected / at risk) | 9/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OROS Hydromorphone (N=20)
Agitation (Psychiatric disorders) | 1
Hypehidrosis (Skin and subcutaneous tissue disorders) | 1
Death due to sepsis (Infections and infestations) | 1
Restlessness (Psychiatric disorders) | 1
Headache (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OROS Hydromorphone (N=20)
Constipation (Gastrointestinal disorders) | 2
Dizziness (Nervous system disorders) | 2
Nausea (Gastrointestinal disorders) | 3
Oedema peripheral (General disorders) | 1
Chest Discomfort (General disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Somnolence (Nervous system disorders) | 1

LIMITATIONS AND CAVEATS:
The study was prematurely terminated due to administrative reason.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No